CLINICAL TRIAL: NCT06645041
Title: The Relationship of Vitamin D and Irisin With Blood Pressure and Heart Rate Variability in Normotensive and Hypertensive Individuals: The Impact of Vitamin D Supplementation in Hypertensive Vitamin D Deficient Patients.
Brief Title: The Impact of Vitamin D Supplementation in Hypertensive Vitamin D Deficient Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sulaimani (Other)
Responsible Party: Principal Investigator, Darya Saeed Abdulateef, Assistant Professor, University of Sulaimani
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CoM-UoS-308
Record Dates: First submitted 2024-10-13; First posted 2024-10-16 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; Vitamin D Deficiency
Keywords: Vitamin D supplementation; Hypertensive vitamin D deficient; Effect on serum Irisin; Effects on HRV
MeSH Terms: conditions — Hypertension; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypertensive Vitamin D deficient individuals receiving placebo capsule (Placebo Comparator): Hypertensive Vitamin D deficient individuals receiving placebo capsules, 1 capsule/week for 8 weeks
  Interventions: Dietary Supplement: Placebo Capsule(s)
- Hypertensive vitamin D deficient individuals receiving Vitamin D supplements (Experimental): Hypertensive Vitamin D deficient individuals receiving Vitamin D capsules, 25,000 IU, 1 capsule/week for 8 weeks
  Interventions: Dietary Supplement: Vitamin D (Cholecalciferol )

INTERVENTIONS:
Dietary Supplement: Vitamin D (Cholecalciferol ) — The hypertensive patients with vitamin D deficiency will receive a Vitamin D capsule with a dose of 25,000 IU. They will be asked to receive a capsule per week for 8 subsequent weeks and re-visit the hospital two weeks from the final dose.
  Arms: Hypertensive vitamin D deficient individuals receiving Vitamin D supplements
Dietary Supplement: Placebo Capsule(s) — The hypertensive patients with vitamin D deficiency will receive a Placebo capsule. They will be asked to receive a capsule per week for 8 subsequent weeks and re-visit the hospital two weeks from the final dose.
  Arms: Hypertensive Vitamin D deficient individuals receiving placebo capsule

SUMMARY:
This study will assess the impact of Vitamin D supplementation on hypertensive patients with Vitamin D deficiency, it will also investigate the relationship between serum Vitamin D, irisin levels, blood pressure, and heart rate variability (HRV) in hypertensive and normotensive individuals.

It is hypothesized that a decrease in blood pressure and an increase in HRV will be noted in the hypertensive treatment group (subjects on supplemental vitamin D) in comparison to the hypertensive control group (placebo) upon vitamin D supplementation.

DETAILED DESCRIPTION:
In a prospective study conducted on 160 participants, 80 hypertensive and 80 normotensive individuals, assessing correlations between Vitamin D, irisin, blood pressure, and HRV, hypertensive vitamin D deficient participants will be recruited in a randomized controlled trial. In this clinical trial, 60 hypertensive participants with Vitamin D deficiency will receive either Vitamin D supplementation (25,000 IU weekly) or a placebo for 8 weeks (30 participants in each group).

Outcome measures include systolic and diastolic blood pressure, HRV, serum Vitamin D, and serum irisin levels before and after supplementation.

The aim is to explore the potential role of Vitamin D and irisin in regulating blood pressure and improving HRV, potentially offering preventive measures for hypertension management.

ELIGIBILITY:
Inclusion Criteria:

Hypertensive: Adult individual diagnosed with hypertension by a specialist (at least two systolic blood pressure readings above 140 mmHg or diastolic blood pressure readings above 90 mmHg, measured by a qualified professional following American Heart Association guidelines) managing hypertension through medication adherence, and regularly attending heart clinic appointments, with no other systemic diseases.

Control: Healthy adult individuals without hypertension or a history of other systemic diseases who volunteer and participate in the study, which will be recruited from relatives, friends, colleagues or patient accompanies. - (*Note: The healthy participants were included in the first part of the study before starting the clinical trial)

Exclusion Criteria:

* 1. Hypertensive individuals who have heart failure and other cardiac or systemic diseases or with recent cardiovascular events.

  2. Secondary hypertension 3. Hypertensive patients who require medication change during the course of the study.

  4. Individuals on Lipid-lowering agents (e.g. simvastatin). 5. The use of other medications affecting blood pressure is not part of the study protocol.

  6. Any subjects on regular supplemental vitamin D or receiving multi-vitamins regularly with vitamin D content of more than 880 IU, one month before recruitment.

  7. Individuals with a BMI over 35 or less than 18 kg/m2. 8. Subjects with a significant change in lifestyle, for example, exercise, weight change, or on a specific dietary regimen during or in the previous four weeks of the study.

  9. Subject diagnosed with neoplasm, or inflammatory or autoimmune diseases 10. Pregnant or lactating female

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-16 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Systolic Blood pressure | 10 weeks
  This measure will track mean changes in systolic blood pressure in mmHg, before and after 8 weeks of Vitamin D supplementation. The objective is to observe whether there is a significant decrease in systolic blood pressure in hypertensive patients receiving Vitamin D compared to those receiving a placebo.
Diastolic Blood pressure | 10 weeks
  This measure will assess mean changes in diastolic blood pressure in mmHg, before and after 8 weeks of Vitamin D supplementation. The study aims to determine if there is a significant decrease in diastolic blood pressure in hypertensive patients receiving Vitamin D compared to the placebo group.
Heart rate variability (HRV) | 10 weeks
  It includes the time domain in milliseconds-ms and frequency domains

SECONDARY OUTCOMES:
Serum Irisin | 10 weeks
  Evaluate changes in mean serum irisin levels in pg/ml or mcg/ml, before and after Vitamin D supplementation in hypertensive patients. The change in mean serum irisin will be correlated with changes in blood pressure and HRV to understand its potential role in cardiovascular regulation.
Serum hydroxycholecalciferol | 10 weeks
  Measure mean serum 25-hydroxyvitamin D levels to confirm the efficacy of supplementation. The levels will be correlated with the mean of blood pressure, HRV, and serum irisin to explore the impact of Vitamin D repletion.

CONTACTS AND LOCATIONS:
Overall Officials: Darya S. Abdulateef, Ph.D., Principal Investigator — University of Sulaimani/College of Medicine/Branch of Medical Education
Locations (3):
- Iraq (3):
  - University of Sulaimani, College of Medicine (CoM-UoS), Sulaymaniyah, Iraq
  - Ministry of Higher Education and Scientific research, University of Sulaimani, College of Medicine (CoM-UoS), Sulaymaniyah, Kurdistan Region
  - Anwar Sheikha Medical City/High quality hospitals, Sulaymaniyah